CLINICAL TRIAL: NCT05118256
Title: An Open, Randomised, Controlled and Unicenter Clinical Trial to Assess the Efficiency of Pirfenidone for the Reduction of Pulmonary Metabolic, Inflammatory and Fibrogenic Activity in Patients With Silicosis Due to Artificial Stone and PMF
Brief Title: Pirfenidone for the Reduction of Metabolic, Inflammatory and Fibrogenic Activity in Complicated Silicosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de investigación e innovación biomédica de Cádiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUN-PIR-2020-01
Record Dates: First submitted 2021-10-01; First posted 2021-11-11 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Silicosis; Progressive Massive Fibrosis; Complicated Silicosis
MeSH Terms: conditions — Silicosis | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Although this is an open study for participants and clinicians, professionals in charge of molecular and cellular analysis, HRCT and PET will be blind to the arm that each subject is assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention - standard of care (No Intervention): A group of patients with PMF will be treated per standard of care on site
- Experimental - Pirfenidone plus standard of care (Experimental): A group of patients with PMF will be treated with pirfenidone plus standard of care on site
  Interventions: Drug: Pirfenidone Oral Tablet

INTERVENTIONS:
Drug: Pirfenidone Oral Tablet — Patients will be treated with pirfenidone (oral tablets) during 6 months
  Other Names: Esbriet
  Arms: Experimental - Pirfenidone plus standard of care

SUMMARY:
Silicosis is one of the leading causes of occupational respiratory disease worldwide. It is due to inhalation of respirable crystalline silica and can lead to progressive massive fibrosis (PMF), respiratory failure, and death. It is estimated that it causes more than 10,000 deaths a year worldwide, mainly in developing countries, although the level of underdiagnosis is high. In developed countries the incidence of the disease has been progressively decreasing in recent years, mainly due to the implementation of effective prevention measures, better occupational health surveillance systems and the displacement of mining activity to other countries, in a way that in the United Kingdom 216 cases were reported from 1996 to 2017. At the moment, there is no curative treatment for the disease, and the only therapeutic option is lung transplantation (when the disease evolves to PMF and subsequent respiratory failure). Meanwhile, the only accepted treatment is supportive treatment, with the administration of oxygen therapy in case of respiratory failure, early treatment of respiratory infections, vaccinations and respiratory rehabilitation. In recent years, molecules with antifibrogenic capacity have been developed and have demonstrated their ability to decrease pulmonary fibrogenic activity in diseases such as Idiopathic Pulmonary Fibrosis (IPF). This has been a milestone in the treatment of this disease and, therefore, its possible application to other diseases that share fibrogenic mechanisms with IPF, as PMF. The two molecules with the most clinical experience and approved for IPF are nintedanib and pirfenidone. The antifibrotic properties of pirfenidone have raised great expectations and many clinical trials are currently being carried out in other lung diseases that cause fibrosis, that is why we decide to study the efficacy of pirfenidone in reducing metabolic, inflammatory, and fibrogenic lung disease in patients with artificial stone silicosis and progressive massive fibrosis (PMF).

DETAILED DESCRIPTION:
Hypothesis: Pirfenidone reduces pulmonary metabolic activity in patients with Progressive Massive Fibrosis (PMF).

Objetives:

Main objetive: To evaluate the efficacy of pirfenidone in reducing pulmonary metabolic activity quantified by PET-CT Scan (F-FDG) in patients with Progressive Massive Fibrosis (PMF).

Secundary objetives:

1. To evaluate the efficacy of pirfenidone in reducing pulmonary inflammatory and fibrogenic activity in patients with Progressive Massive Fibrosis (PMF), quantified by cell biomarkers, and the relation with the pulmonary metabolic activity.
2. To assess changes brought about by pirfenidone in the different cells biomarkers patterns and metabolic activity resulted by PET/TC with 18-FDG
3. To assess radiological changes in HRCT (High Resolution Computed Tomography) that occur after administration of pirfenidone and the relation with biomarkers and with 18F FDG acquisition.
4. To assess wheter administration of pirfenidone generates changes on standard funtional respiratory explorations, and the relation with inflammatory and metabolic activity. 5. To assess clinical changes (if any) and safety of pirfenidone after administration to patients with PMF.

Methodology: An Open, Randomised, Controlled, 2 arms and Unicenter Clinical Trial to Assess the Efficiency of Pirfenidone for the Reduction of Pulmonary Metabolic, Inflammatory and Fibrogenic Activity in Patients With Silicosis Due to Artificial Stone and PMF.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age over 18 years and under 65.
* 2. Man with a diagnosis of silicosis in the form of PMF by lung or lymph node biopsy, or by radiological criteria.
* 3. History of exposure to silica in work with artificial stone for at least 5 years.
* 4. Patients capable of consenting to their participation in the study by providing written informed consent, or, if they are not trained, through a legal repressentative.

Exclusion Criteria:

* 1. Participation in another clinical trial in the 6 months prior to the start of participation in this study.
* 2. Hypersensitivity to any of the components of pirfenidone.
* 3. Biological or farmacological treatment for any other disease or condition related to silicosis or PMF. Exception: prednisona (or equivalent) dose 20mg per day or lower.
* 4. Concomitant treatment with a drug that can causes pirfenidone interactions: Cytotoxic drugs, immunosuppressants, cytokine modulators including but not limited to azathioprine, bosentan, ambrisentan, cyclophosphramide, cyclosporine, etarnecept, iloprost, infliximab, leukotriene antagonists, methotrexate, mycophenolate , tacrolimus, montelukast, tetrathiomolybdate, TNF-alpha inhibitors, imatinib mesylate, interferon gamma 1-beta, and tyrosine kinase inhibitors. Strong CYP1A2 inhibitors (eg fluvoxamine, enoxacin), P-glycoprotein or CYP3A4 inhibitors (eg Ketoconazole, erythromycin), or their inducers (eg rifampicin, carbamazepine, phenytoin). Other moderate CYP1A2 inhibitors (eg amiodarone or propafenone) which will also be prohibited. Any investigational therapy in an active clinical trial. Grapefruit juice.
* 5. Active infectious disease.
* 6. Any pathology that may condition the evolution of respiratory diseases, including cancer, HIV, HBV, HCV, liver cirrhosis, liver failure, severe kidney failure or any other that in the opinion of the investigator may interfere with the results of the study.
* 7. Active smoking.
* 8. Laboratory test abnormalities at screening timepoint - Total bilirrubin >2 ULN - AST/SGOT or ALT/SGPT > 2.5 ULN - Alkaline phosphatase >3.0 ULN - Creatinine clearance <40 mL/min (Cockcroft-Gault).
* 9. Concomitant treatments that may cause serious digestive events.
* 10. Digestive surgery or similar procedures that may cause digestive intolerances.
* 11. Not availability to complete all the trial visits.
* 12. Angiodema

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-11-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Metabolic pulmonary activity assessed by PET-CT Scan (18 FFDG) | baseline (day 1), month 6, month 12
  Metabolic pulmonary activity assessed by PET-CT Scan (18 FFDG) in patients treated with pirfenidone vs control patients. The variables will be analyzed in lung and mediastinum independently and the measurement of the metabolic response will be based on the standardized uptake value (SUV) at its maximum (SUVmax) and mean (SUVmean) values.

SECONDARY OUTCOMES:
Cell biomarkers in peripheral blood: - Pro/anti fibrotic and pro/anti inflammatory biomarkers | baseline (day 1), month 3, month 6, month 9, month 12
  Pro/anti fibrotic and pro/anti inflammatory biomarkers: cytokines (IL-1α, IL-1β, IL-1RA, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12 (p40), IL-12 (p70), IL-13, IL-15, IL-17, IL-18, IP-10, TGF-β, TNF-α, IFN-γ, MIP-1α, MIP-1β, MCP-1, PDGF, bFGF, MMP1, -2, -7, -9, -10). Immunological biomarkers: CD45, CD45RO, CD45RA, CD3, CD4, CD8, CD19, CD27, CD56, CD126, CD25, INF-γ, IL-4, FoxP3, CD196 y CD161 Note: There are no previous studies in patients with artificial stone silicosis in which they have analyzed the indicated biomarkers. This is a comprehensive preliminary analysis of biomarkers and we want to correlate the obtained values with the results derived from PET-CT in both groups of patients in the trial.
Number of adverse events (AE) and adverse reactions (AR), of serious adverse events (SAE) and serious and unexpected adverse reactions (SUSAR). | baseline (day 1), month 3, month 6, month 9, month 12
  Number of adverse events (AE) and adverse reactions (AR), of serious adverse events (SAE) and serious and unexpected adverse reactions (SUSAR).
Respiratory symptoms (cough, expectoration and dyspnea) and quality of life related to health using the EQ-5D 5L test. | baseline (day 1), month 3, month 6, month 9, month 12
  Respiratory symptoms (cough, expectoration and dyspnea) and quality of life related to health using the EQ-5D 5L test.
Respiratory function variables | baseline (day 1), month 3, month 6, month 9 and month 12
  Forced Vital Capacity (FVC), Forced Expiratory Volume in the first second, ratio Forced Expiratory in the first second / Forced Vital Capacity and Diffusing Capacity of the lungs for carbon monoxide, obtained through standardized respiratory function tests.
Radiological categorization by chest radiology and by High Resolution Computed Tomography, following the International Classification of High-resolution Computed Tomography for Occupational and Environmental Respiratory Diseases (ICOERD) | baseline (day 1), month 6, month 12
  Radiological categorization by chest radiology and by High Resolution Computed Tomography, following the International Classification of High-resolution Computed Tomography for Occupational and Environmental Respiratory Diseases (ICOERD)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio León Jiménez, MD, Principal Investigator — Fundación Cádiz- INIBICA; Antonio Campos Caro, phD, Principal Investigator — Fundación Cádiz- INIBICA
Locations (1):
- Antonio León Jiménez, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No
The study results will be published in scientific pneumologic journal and available in PubMed and clinicaltrials website